CLINICAL TRIAL: NCT01741805
Title: The Clinical and Laboratory Phenotypes of Severe Asthma Patients in Clalit Health Services Haifa.
Status: Withdrawn | Type: Observational
Why Stopped: Slow recruitment of patients
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-12-0032-CTIL
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe Asthma: Patients with severe asthma as specified under inclusion, exclusion criteria
  Interventions: Other: Severe Asthma

INTERVENTIONS:
Other: Severe Asthma — Demographic data, Spirometry, induced sputum, IgE, Aspergillus specific IgE

SUMMARY:
Asthma is a chronic illness characterized by inflammation of the airways. Severe asthma is defined in the literature as asthma not controlled by medication. In recent years it has become known that severe asthma is a variable disease and has subtypes relating to the age of onset, type of inflammation and allergy, obesity, etc.

Our aim is to characterize the phenotypes of severe asthma population in our clinic and compare the prevalent phenotypes to the phenotypes described before.

DETAILED DESCRIPTION:
Study measures will include the following:

* asthma demographic and symptoms questionnaire
* Validation of proper inhaler technique
* Height, weight measurements
* Forced spirometry and reversibility testing
* DLCO
* Fractional excretion of NO in exhaled breath
* Chest and sinus CT
* Induced sputum analysis
* Complete blood count, electrolytes, immunoglobulin E, Aspergillus Specific IgE
* Skin allergy testing

ELIGIBILITY:
Inclusion Criteria:

1. Presence of Asthma- typical symptoms and signs accompanied by either: a. obstruction in Spirometry, OR- b. positive methacholine test
2. Regular use of high dose of inhaled corticosteroids (1000 micrograms of fluticasone per day or equivalent) in addition to a long acting beta agonist (LABA).
3. Lack of asthma control- 2 or more exacerbations in the past year- exacerbations defined by hospitalization or care in an emergency department or treatment with systemic glucocorticosteroids for exacerbation of asthma symptoms.

Exclusion Criteria:

1. Presence of another relevant respiratory illness, such as chronic obstructive pulmonary disease (COPD)
2. lack of adherence to medical therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of petients with severe asthma, described by presence of symptoms despite adequate treatment as described in the following sections.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 1 year

SECONDARY OUTCOMES:
Carbon Monoxide Diffusion Capacity (DLCO) | 1 year
Percent eosinophils in induced sputum sample | 1 year
Bronchiectasis on computerized tomography (CT) | 1 year)
Blood level of Total immunoglobulin E (IgE) | 1 year
Presence of blood antibody to Aspergillus Fumigatus | 1 year
Fraction of Nitric Oxide (NO) in expired air | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michal Shteinberg, MD,PhD, Principal Investigator — Pulmonology Institute, Carmel Medical Center
Locations (1):
- Pulmonology Institute, Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No